CLINICAL TRIAL: NCT05705167
Title: A Multicentre, Open Label, Randomised, Controlled, Basket, Pragmatic, Phase II, Clinical and Translational Study to Determine the Efficacy and Safety of Plitidepsin Versus Control in Immunocompromised Adult Patients With Symptomatic COVID-19 Requiring Hospital Care
Brief Title: Plitidepsin Versus Control in Immunocompromised Adult Participants With Symptomatic COVID-19 Requiring Hospital Care (NEREIDA)
Acronym: NEREIDA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Significant difficulties in the recruitment of participants.
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AV-APL-B-002-22; 2022-002489-34 (EudraCT Number)
Record Dates: First submitted 2022-12-21; First posted 2023-01-30 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: COVID-19; Plitidepsin
MeSH Terms: conditions — COVID-19 | interventions — plitidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plitidepsin 2.5 mg (Experimental): Best standard care (as per applicable local, institutional, national, supranational COVID-19 treatment guidelines) and plitidepsin (administered as a 60-minute intravenous (IV) infusion, every 24 hours for 3 consecutive days, at a dose of 2.5 mg) will be administered to participants of the following groups:
  * Group 1 - Participants receiving immune-suppression due to haematopoietic or organ transplantation.
  * Group 2 - Participants receiving B-cell depleting therapies.
  * Group 3 - Participants receiving other immune-suppressive therapies.
  * Group 4 - Other situations with immune deficiencies.
  Interventions: Drug: Plitidepsin
- Control (No Intervention): Best standard care (as per applicable local, institutional, national, supranational COVID-19 treatment guidelines) ± other regulatory-approved antiviral (if clinically indicated) will be administered to participants of the following groups:
  * Group 1 - Participants receiving immune-suppression due to haematopoietic or organ transplantation.
  * Group 2 - Participants receiving B-cell depleting therapies.
  * Group 3 - Participants receiving other immune-suppressive therapies.

INTERVENTIONS:
Drug: Plitidepsin — IV infusion over 60-minutes
  Arms: Plitidepsin 2.5 mg

SUMMARY:
The primary objective of this study is to evaluate efficacy of plitidepsin in pre-specified groups of immunocompromised patients with symptomatic COVID-19 requiring hospital care versus control in terms of mortality.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to initiation of any study-specific procedures and study treatment.
* Participant aged ≥18 years.
* Participant diagnosed COVID-19, with the following characteristics:

  1. A regulatory-approved test, collected no more than 3 days prior to study randomisation, with either a Ct value ≤30 or a positive antigen test.
  2. Presence of any of the selected signs/symptom listed in the COVID-19 signs/symptoms checklist within the last 24 hours.
* Participant already admitted or requiring hospital care for symptomatic COVID-19, for which at least one antiviral has failed or cannot be used (i.e., contraindication, absence of labelled indication, guidelines or drug unavailability), after a minimum washout period of 24 hours for small molecules (e.g., remdesivir, molnupiravir, nirmaltrevir, ritonavir) and 5 days for antiviral monoclonal antibodies (e.g., tixagevimab + cilgavimab) or convalescent plasma.
* Adequate bone marrow, liver, kidney, and metabolic function, defined by the following tests performed at local laboratory:

  1. Absolute neutrophil count ≥500/mm^3 (0.5 x 109/L).
  2. Platelet count ≥ 50 000/mm3 (50 x 109/L).
  3. Alanine transaminase (ALT) ≤3 x upper limit of normal (ULN) (≤5 x ULN if preexistent liver involvement by the underlying disease).
  4. Serum bilirubin ≤1.5 x ULN (or direct bilirubin <1.5 x ULN when total bilirubin is above ULN).
  5. Estimated glomerular filtration rate ≥30 mL/min (CKD-EPI Creatinine Equation [2021]).
* Females of child-bearing potential must have a negative serum or urine pregnancy test by local laboratory at screening and must be non-lactating.
* Females of child-bearing potential and fertile males with partners of child-bearing potential must use contraceptive methods as specified in the protocol.

Group-specific inclusion criteria:

* Group 1 - Patients receiving, within the last 30 days, immune-suppressive therapy due to haematopoietic or organ transplantation.
* Group 2 - Participants receiving B-cell depleting therapies within the last 6 months (with the exception of CAR-T cell therapy for which time restriction is not applicable).
* Group 3 - Participants receiving, within the last 30 days, other immune-suppressive therapies.
* Group 4 - Other situations with immunodeficiency.

  1. Primary immune deficiencies.
  2. Human immunodeficiency virus (HIV) infection, with CD4^+ T lymphocyte < 200 cells/μL in the last month.
  3. Radiation therapy within the last 3 months- requires documentation of ALC < 500 cells/μL.
  4. Haematological neoplasia or myelodysplasia not currently receiving any therapy.
  5. Other situations with a documentation of ALC < 500 cells/μL.

Exclusion Criteria:

* Evidence of critical illness.
* Any of the following cardiac conditions or risk factors:

  1. Cardiac infarction or cardiac surgery episode within the last month.
  2. History of known congenital QT prolongation.
  3. Known structural cardiomyopathy with abnormal left ventricular ejection fraction (LVEF) (<50%).
  4. Current clinical evidence of heart failure or acute cardiac ischaemia (New York Heart Association (NYHA) class III-IV).
* Hypersensitivity to the active ingredient or any of the excipients (mannitol, macrogolglycerol hydroxystearate, and ethanol) or contraindication to receive dexamethasone, antihistamine H1/H2, or anti-serotoninergic 5HT3 agents.
* Females who are pregnant or breast-feeding.
* Females and males with partners of child-bearing potential who are not using at least 1 protocol-specified method of contraception.
* Any situation currently requiring increasing needs of immune-suppressive agents.
* Any other clinically significant medical condition or laboratory abnormality that, in the opinion of the investigator, would jeopardise the safety of the participant or potentially impact on participant compliance or the safety/efficacy observations in the study.
* Participation in another clinical study involving an investigational drug within 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Flemish Brabant, Belgium
- France (5):
  - Cancer Research Centre of Lyon, Lyon, Auvergne-Rhône-Alpes
  - Hôpitaux Civils de Colmar - Centre Hospitalier Louis Pasteur, Colmar, Grand Est
  - Centre Hospitalier Régional Universitaire de Tours, Tours, Indre-et-Loire
  - Centre Hospitalier de la Côte Basque, Bayonne, Pyrénées-Atlantiques
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
- Georgia (3):
  - The First University Clinic of the Tbilisi State Medical University, Tbilisi
  - Ltd Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Tbilisi
  - Academician Vakhtang Bochorishvili Clinic, Tbilisi
- Greece (6):
  - General Hospital of Athens Evangelismos, Athens, Attica
  - Laiko General Hospital of Athens, Athens, Attica
  - Alexandra General Hospital, Athens, Attica
  - University General Hospital Attikon, Athens, Attica
  - University Hospital of Ioannina, Ioannina, Epirus
  - General Hospital for Thoracic Diseases Sotiria, Athens
- Országos Korányi Pulmonológiai Intézet, Budapest, Hungary
- Sheba Medical Center Hospital - Tel Hashomer, Ramat Gan, Tel Aviv, Israel
- Italy (2):
  - IRCCS Istituto Nazionale per le Malattie Infettive Lazzaro Spallanzani, Roma, Rome
  - Ente Ospedaliero Ospedali Galliera, Genova
- Wojewódzki Specjalistyczny Szpital im. Dr. Władysława Biegańskiego, Lodz, Lódzkie, Poland
- Portugal (4):
  - Hospital da Senhora da Oliveira - Guimarães, Guimarães, Braga District
  - Centro Hospitalar Universitário Lisboa Norte, E.P.E - Hospital De Santa Maria, Lisbon, Lisbon District
  - Hospital Pedro Hispano, Senhora da Hora
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, Vila Nova de Gaia
- Spain (18):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Alvaro Cunqueiro - Clinico Universitario Vigo, Vigo, Pontevedra
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - Vall d'Hebron Institut de Recerca, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Regional Universitario de Málaga - Hospital General, Málaga
  - Complejo Asistencial Universitario de Salamanca - Hospital Clínico, Salamanca
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (2):
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, England
  - University College London Hospitals NHS Foundation Trust, London

REFERENCES:
- [Derived] Landete P, Caliman-Sturdza OA, Lopez-Martin JA, Preotescu L, Luca MC, Kotanidou A, Villares P, Iglesias SP, Guisado-Vasco P, Saiz-Lou EM, Del Carmen Farinas-Alvarez M, de Lucas EM, Perez-Alba E, Cisneros JM, Estrada V, Hidalgo-Tenorio C, Poulakou G, Torralba M, Fortun J, Garcia-Ocana P, Lemaignen A, Marcos-Martin M, Molina M, Paredes R, Perez-Rodriguez MT, Raev D, Ryan P, Meira F, Gomez J, Torres N, Lopez-Mendoza D, Jimeno J, Varona JF. A Phase III Randomized Controlled Trial of Plitidepsin, a Marine-Derived Compound, in Hospitalized Adults With Moderate COVID-19. Clin Infect Dis. 2024 Oct 15;79(4):910-919. doi: 10.1093/cid/ciae227. PMID 39182994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 37 participants were enrolled at 15 investigative sites between April 2023 and April 2024. Randomised participants who received at least 1 dose of study treatment and completed follow-up for survival until Day 30 (±2) were included in the Full Analysis Set (FAS) population.
Groups:
- Group 1: Plitidepsin 2.5 mg: Best standard care (as per applicable local, institutional, national, supranational COVID-19 treatment guidelines) and plitidepsin (administered as a 60-minute intravenous (IV) infusion, every 24 hours for 3 consecutive days, at a dose of 2.5 mg) were administered to participants in Group 1.
  Group 1 - Participants who received immune-suppression due to haematopoietic or organ transplantation.
- Group 1: Control: Best standard care (as per applicable local, institutional, national, supranational COVID-19 treatment guidelines) ± other regulatory-approved antiviral (if clinically indicated) were administered to participants in Group 1.
  Group 1 - Participants who received immune-suppression due to haematopoietic or organ transplantation.
- Group 2: Plitidepsin 2.5 mg: Best standard care (as per applicable local, institutional, national, supranational COVID-19 treatment guidelines) and plitidepsin (administered as a 60-minute IV infusion, every 24 hours for 3 consecutive days, at a dose of 2.5 mg) were administered to participants in Group 2.
  Group 2 - Participants who received B-cell depleting therapies.
- Group 2: Control: Best standard care (as per applicable local, institutional, national, supranational COVID-19 treatment guidelines) ± other regulatory-approved antiviral (if clinically indicated) were administered to participants in Group 2.
  Group 2 - Participants who received B-cell depleting therapies.
- Group 3: Plitidepsin 2.5 mg: Best standard care (as per applicable local, institutional, national, supranational COVID-19 treatment guidelines) and plitidepsin (administered as a 60-minute IV infusion, every 24 hours for 3 consecutive days, at a dose of 2.5 mg) were administered to participants in Group 3.
  Group 3 - Participants who received other immune-suppressive therapies.
- Group 3: Control: Best standard care (as per applicable local, institutional, national, supranational COVID-19 treatment guidelines) ± other regulatory-approved antiviral (if clinically indicated) were administered to participants in Group 3.
  Group 3 - Participants who received other immune-suppressive therapies.
- Group 4: Plitidepsin 2.5 mg: Best standard care (as per applicable local, institutional, national, supranational COVID-19 treatment guidelines) and plitidepsin (administered as a 60-minute IV infusion, every 24 hours for 3 consecutive days, at a dose of 2.5 mg) were administered to participants in Group 4.
  Group 4 - Other situations with immune deficiencies.
Period: Overall Study
Arm/Group | Group 1: Plitidepsin 2.5 mg | Group 1: Control | Group 2: Plitidepsin 2.5 mg | Group 2: Control | Group 3: Plitidepsin 2.5 mg | Group 3: Control | Group 4: Plitidepsin 2.5 mg
Started | 2 | 3 | 11 | 11 | 1 | 1 | 8
Completed | 2 | 1 | 7 | 3 | 0 | 0 | 6
Not Completed | 0 | 2 | 4 | 8 | 1 | 1 | 2
Not completed — Randomised but not Treated | 0 | 2 | 0 | 7 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 3 | 0 | 1 | 1 | 1
Not completed — Discontinued Prior to FAS Eligibility | 0 | 0 | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: FAS Population: All randomised participants who received at least 1 dose of study treatment (plitidepsin or control) and completed follow-up for survival until Day 30 (±2). Participants who died before the end of the follow-up period were also included in the FAS population.
Groups:
- Group 1: Plitidepsin 2.5 mg: Best standard care (as per applicable local, institutional, national, supranational COVID-19 treatment guidelines) and plitidepsin (administered as a 60-minute IV infusion, every 24 hours for 3 consecutive days, at a dose of 2.5 mg) were administered to participants in Group 1.
  Group 1 - Participants who received immune-suppression due to haematopoietic or organ transplantation.
- Total: Total of all reporting groups
Arm/Group | Group 1: Plitidepsin 2.5 mg | Group 1: Control | Group 2: Plitidepsin 2.5 mg | Group 2: Control | Group 3: Plitidepsin 2.5 mg | Group 3: Control | Group 4: Plitidepsin 2.5 mg | Total
Number analyzed (Participants) | 2 | 1 | 10 | 3 | 1 | 1 | 7 | 25
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 6
  ≥ 65 years - < 75 years | 1 | 1 | 6 | 2 | 0 | 1 | 1 | 12
  ≥ 75 years | 0 | 0 | 1 | 0 | 1 | 0 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 5 | 2 | 0 | 0 | 5 | 14
  Male | 1 | 0 | 5 | 1 | 1 | 1 | 2 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 2 | 1 | 10 | 3 | 1 | 1 | 5 | 23
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Ethnicity was not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: One-month All-cause Mortality Rate
Description: In the event of the participant initiating another non-protocol therapy, 1-month all-cause mortality rate was evaluated regardless of initiation of new non-protocol therapy.
Time Frame: Day 1 to Day 30 (±2)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Plitidepsin 2.5 mg | Group 1: Control | Group 2: Plitidepsin 2.5 mg | Group 2: Control | Group 3: Plitidepsin 2.5 mg | Group 3: Control | Group 4: Plitidepsin 2.5 mg
Number analyzed (Participants) | 2 | 1 | 10 | 3 | 1 | 1 | 7
percentage of participants | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 97.5] | 20.0 [2.5 to 55.6] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 97.5] | 100.0 [2.5 to 100.0] | 14.3 [0.4 to 57.9]

2. Secondary Outcome: Time to Confirmed Negativisation in SARS-CoV-2 Antigen Test or Real Time Polymerase Chain Reaction (RT-PCR) Cycle Threshold (Ct) > 30
Description: Time to confirmed negativisation in SARS-CoV antigen test or RT-PCR Ct>30 was calculated as time from randomisation to the corresponding event using Kaplan-Meier (KM) estimates. Participants with no available data for any time to event efficacy endpoint were censored at time 0, end of study (Day 60 ±3), or date of early study termination. Also, participants who had not achieved the time to event endpoint were censored at the last valid assessment.
Time Frame: Day 1 to Day 60 (±3)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Group 1: Plitidepsin 2.5 mg | Group 1: Control | Group 2: Plitidepsin 2.5 mg | Group 2: Control | Group 3: Plitidepsin 2.5 mg | Group 3: Control | Group 4: Plitidepsin 2.5 mg
Number analyzed (Participants) | 2 | 1 | 10 | 3 | 1 | 1 | 7
days | 61.0 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 2.0 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 14.0 [2.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 14.0 [4.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 13.0 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 10.0 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 14.0 [3.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median.

3. Secondary Outcome: Time to Sustained End of COVID-related Hospital Care
Description: Time to sustained end of COVID-related hospital care from the time of randomisation was calculated as time from randomisation to the corresponding event using KM estimates. Participants with no available data for any time to event efficacy endpoint were censored at time 0, end of study (Day 60 ±3), or date of early study termination. Also, participants who had not achieved the time to event endpoint were censored at the last valid assessment.
Time Frame: Day 1 to Day 60 (±3)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Group 1: Plitidepsin 2.5 mg | Group 1: Control | Group 2: Plitidepsin 2.5 mg | Group 2: Control | Group 3: Plitidepsin 2.5 mg | Group 3: Control | Group 4: Plitidepsin 2.5 mg
Number analyzed (Participants) | 2 | 1 | 10 | 3 | 1 | 1 | 7
days | 20.5 [2.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 4.0 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 4.5 [2.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 37.0 [13.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 24.0 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 2.0 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 7.0 [3.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median.

4. Secondary Outcome: Time to Sustained Improvement and Resolution of Selected COVID-19 Signs/Symptoms
Description: Time to sustained improvement and resolution of all targeted COVID-19 signs/symptoms was calculated as time from randomisation to the corresponding event using KM estimates. Corresponding events were defined as the event occurring on the first of 4 consecutive days when all symptoms scored as National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v5.0; category of moderate-severe intensity, or requiring medical intervention, or limiting instrumental activity of daily living are scored as mild or absent AND all symptoms scored mild or 0 (absent) at study entry are scored as 0. Participants with no available data for any time to event efficacy endpoint were censored at time 0, end of study (Day 60 ±3), or date of early study termination. Also, participants who had not achieved the time to event endpoint were censored at the last valid assessment.
Time Frame: Day 1 to Day 60 (±3)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Group 1: Plitidepsin 2.5 mg | Group 1: Control | Group 2: Plitidepsin 2.5 mg | Group 2: Control | Group 3: Plitidepsin 2.5 mg | Group 3: Control | Group 4: Plitidepsin 2.5 mg
Number analyzed (Participants) | 2 | 1 | 10 | 3 | 1 | 1 | 7
days | NA [5.0 to NA] — Median and upper confidence interval were not calculable due to fewer than 50% events. | NA [NA to NA] — Median and confidence intervals were not calculable due to insufficient event data. | NA [3.0 to NA] — Median and upper confidence interval were not calculable due to fewer than 50% events. | 14.0 [4.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 17.0 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 2.0 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 37.0 [2.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median.

5. Secondary Outcome: Number of Participants in Each Category of the World Health Organization (WHO) Clinical Progression Scale (CPS)
Description: Distribution of participants according to their clinical status by the 11-category WHO CPS:
  * Uninfected; no viral ribonucleic acid (RNA) detected
  * Asymptomatic; viral RNA detected
  * Symptomatic; independent
  * Symptomatic; assistance needed
  * Hospitalised; no oxygen therapy
  * Hospitalised; oxygen by mask or nasal prongs
  * Hospitalised; oxygen by non-invasive ventilation (NIV) or high flow
  * Intubation and mechanical ventilation
  * Mechanical ventilation or vasopressors
  * Mechanical ventilation and vasopressors, dialysis, or extracorporeal membrane oxygenation (ECMO) OR
  * Death.
Time Frame: Days 4 (±1), 8 (±1), 15 (±1), 30 (±2), and 60 (±3)
Population: FAS Population: All randomised participants who received at least 1 dose of study treatment (plitidepsin or control) and completed follow-up for survival until Day 30 (±2). Participants who died before the end of the follow-up period were also included in the FAS population. Number of participants analysed represents participants with available data at each individual timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Plitidepsin 2.5 mg | Group 1: Control | Group 2: Plitidepsin 2.5 mg | Group 2: Control | Group 3: Plitidepsin 2.5 mg | Group 3: Control | Group 4: Plitidepsin 2.5 mg
Number analyzed (Participants) | 2 | 1 | 10 | 3 | 1 | 1 | 7
Participants
  Day 4: number analyzed (Participants) | 2 | 1 | 9 | 3 | 1 | 0 | 7
  Day 4: Uninfected; no viral RNA detected | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 4: Asymptomatic; viral RNA detected | 0 | 0 | 2 | 0 | 0 |  | 0
  Day 4: Symptomatic; independent | 1 | 0 | 1 | 0 | 0 |  | 0
  Day 4: Symptomatic; assistance needed | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 4: Hospitalised; no oxygen therapy | 0 | 1 | 4 | 2 | 0 |  | 5
  Day 4: Hospitalised; oxygen by mask or nasal prongs | 1 | 0 | 0 | 1 | 0 |  | 1
  Day 4: Hospitalised; oxygen by NIV or high flow | 0 | 0 | 2 | 0 | 1 |  | 1
  Day 4: Intubation and mechanical ventilation | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 4: Mechanical ventilation or vasopressors | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 4: Mechanical ventilation and vasopressors, dialysis, or ECMO | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 4: Dead | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 8: Uninfected; no viral RNA detected | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Day 8: Asymptomatic; viral RNA detected | 0 | 0 | 3 | 0 | 0 | 0 | 2
  Day 8: Symptomatic; independent | 1 | 0 | 4 | 1 | 0 | 0 | 1
  Day 8: Symptomatic; assistance needed | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8: Hospitalised; no oxygen therapy | 0 | 0 | 0 | 2 | 0 | 0 | 1
  Day 8: Hospitalised; oxygen by mask or nasal prongs | 1 | 0 | 1 | 0 | 0 | 0 | 1
  Day 8: Hospitalised; oxygen by NIV or high flow | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Day 8: Intubation and mechanical ventilation | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8: Mechanical ventilation or vasopressors | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Day 8: Mechanical ventilation and vasopressors, dialysis, or ECMO | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8: Dead | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 15: number analyzed (Participants) | 2 | 1 | 10 | 3 | 1 | 1 | 6
  Day 15: Uninfected; no viral RNA detected | 0 | 1 | 2 | 0 | 0 | 1 | 1
  Day 15: Asymptomatic; viral RNA detected | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Day 15: Symptomatic; independent | 1 | 0 | 1 | 1 | 0 | 0 | 1
  Day 15: Symptomatic; assistance needed | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Day 15: Hospitalised; no oxygen therapy | 1 | 0 | 1 | 1 | 0 | 0 | 1
  Day 15: Hospitalised; oxygen by mask or nasal prongs | 0 | 0 | 0 | 1 | 1 | 0 | 1
  Day 15: Hospitalised; oxygen by NIV or high flow | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 15: Intubation and mechanical ventilation | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 15: Mechanical ventilation or vasopressors | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Day 15: Mechanical ventilation and vasopressors, dialysis, or ECMO | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Day 15: Dead | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 30: number analyzed (Participants) | 2 | 1 | 7 | 3 | 1 | 0 | 5
  Day 30: Uninfected; no viral RNA detected | 0 | 1 | 3 | 1 | 0 |  | 2
  Day 30: Asymptomatic; viral RNA detected | 0 | 0 | 2 | 0 | 0 |  | 2
  Day 30: Symptomatic; independent | 2 | 0 | 1 | 0 | 0 |  | 0
  Day 30: Symptomatic; assistance needed | 0 | 0 | 0 | 0 | 1 |  | 1
  Day 30: Hospitalised; no oxygen therapy | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 30: Hospitalised; oxygen by mask or nasal prongs | 0 | 0 | 0 | 2 | 0 |  | 0
  Day 30: Hospitalised; oxygen by NIV or high flow | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 30: Intubation and mechanical ventilation | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 30: Mechanical ventilation or vasopressors | 0 | 0 | 1 | 0 | 0 |  | 0
  Day 30: Mechanical ventilation and vasopressors, dialysis, or ECMO | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 30: Dead | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 60: number analyzed (Participants) | 2 | 1 | 6 | 3 | 1 | 0 | 5
  Day 60: Uninfected; no viral RNA detected | 1 | 1 | 3 | 1 | 0 |  | 4
  Day 60: Asymptomatic; viral RNA detected | 1 | 0 | 2 | 1 | 0 |  | 0
  Day 60: Symptomatic; independent | 0 | 0 | 1 | 0 | 0 |  | 1
  Day 60: Symptomatic; assistance needed | 0 | 0 | 0 | 0 | 1 |  | 0
  Day 60: Hospitalised; no oxygen therapy | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 60: Hospitalised; oxygen by mask or nasal prongs | 0 | 0 | 0 | 1 | 0 |  | 0
  Day 60: Hospitalised; oxygen by NIV or high flow | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 60: Intubation and mechanical ventilation | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 60: Mechanical ventilation or vasopressors | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 60: Mechanical ventilation and vasopressors, dialysis, or ECMO | 0 | 0 | 0 | 0 | 0 |  | 0
  Day 60: Dead | 0 | 0 | 0 | 0 | 0 |  | 0

6. Secondary Outcome: Number of Participants Requiring Oxygen Therapy
Description: The maximum number of participants requiring oxygen therapy on any day during each visit window is reported.
Time Frame: Days 4 (±1), 8 (±1), 15 (±1), 30 (±2), and 60 (±3)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Plitidepsin 2.5 mg | Group 1: Control | Group 2: Plitidepsin 2.5 mg | Group 2: Control | Group 3: Plitidepsin 2.5 mg | Group 3: Control | Group 4: Plitidepsin 2.5 mg
Number analyzed (Participants) | 2 | 1 | 10 | 3 | 1 | 1 | 7
Participants
  Day 4 | 0 | 0 | 2 | 1 | 1 | 0 | 3
  Day 8 | 1 | 0 | 3 | 1 | 1 | 0 | 3
  Day 15 | 0 | 0 | 3 | 1 | 1 | 1 | 1
  Day 30 | 0 | 0 | 1 | 1 | 1 | 0 | 1
  Day 60 | 0 | 0 | 1 | 1 | 0 | 0 | 0

7. Secondary Outcome: Time to Sustained Discontinuation of Oxygen Supplementation
Description: Time to sustained discontinuation is calculated as time from randomisation to the corresponding event using KM estimates. Corresponding events were defined as discontinuation of oxygen supplementation for at least 7 days. Participants with no available data for any time to event efficacy endpoint were censored at time 0, end of study (Day 60 ±3), or date of early study termination. Also, participants who had not achieved the time to event endpoint were censored at the last valid assessment.
Time Frame: Day 1 to Day 60 (±3)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Group 1: Plitidepsin 2.5 mg | Group 1: Control | Group 2: Plitidepsin 2.5 mg | Group 2: Control | Group 3: Plitidepsin 2.5 mg | Group 3: Control | Group 4: Plitidepsin 2.5 mg
Number analyzed (Participants) | 2 | 1 | 10 | 3 | 1 | 1 | 7
days | 13.0 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | NA [NA to NA] — Median and confidence intervals were not calculable due to insufficient event data occurring. | 63.0 [1.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | NA [34.0 to NA] — Median and upper confidence interval were not calculable due to fewer than 50% events. | NA [NA to NA] — Median and confidence intervals were not calculable due to insufficient event data occurring below the median. | 14.0 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 14.0 [2.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median.

8. Secondary Outcome: Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE)
Description: Frequency of the following events (all-cause and treatment-related) are included:
  * TEAEs
  * TEAEs ≥ grade 3 according to the NCI CTCAE v5.0
  * TEAEs of special interest
  * Serious TEAEs
  * Serious adverse reactions (SARs)
  * AEs leading to treatment discontinuation
  * Deaths (related to COVID-19/all)
  Clinically relevant/significant changes from Baseline in laboratory parameters and vital signs were reported as AEs.
Time Frame: Day 1 to Day 60 (±3)
Population: As Treated Population: All participants who received any exposure to study treatment (plitidepsin or control). As Treated population was analysed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Plitidepsin 2.5 mg | Group 1: Control | Group 2: Plitidepsin 2.5 mg | Group 2: Control | Group 3: Plitidepsin 2.5 mg | Group 3: Control | Group 4: Plitidepsin 2.5 mg
Number analyzed (Participants) | 2 | 1 | 11 | 4 | 1 | 1 | 8
Participants
  Any TEAE | 1 | 1 | 10 | 4 | 1 | 1 | 7
  Any treatment-related TEAE | 1 | 0 | 4 | 1 | 0 | 0 | 2
  Any TEAE ≥ grade 3 | 1 | 0 | 5 | 4 | 1 | 1 | 4
  Any treatment-related TEAE ≥ grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Any TEAE of special interest | 1 | 0 | 4 | 2 | 0 | 0 | 4
  Any treatment-related TEAE of special interest | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Any serious TEAE | 1 | 0 | 5 | 4 | 1 | 1 | 2
  Any treatment-related serious TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to treatment discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any treatment-related TEAE leading to treatment discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to death | 0 | 0 | 3 | 0 | 1 | 1 | 1
  Any treatment-related TEAE leading to death | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 60 (±3)
Description: As Treated Population: All participants who received any exposure to study treatment (plitidepsin or control). As Treated population was analysed according to the treatment they actually received.
Arm/Group | Group 1: Plitidepsin 2.5 mg | Group 1: Control | Group 2: Plitidepsin 2.5 mg | Group 2: Control | Group 3: Plitidepsin 2.5 mg | Group 3: Control | Group 4: Plitidepsin 2.5 mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 3/11 | 0/4 | 1/1 | 1/1 | 1/8
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1 | 5/11 | 4/4 | 1/1 | 1/1 | 2/8
Other Adverse Events (participants affected / at risk) | 1/2 | 1/1 | 10/11 | 4/4 | 1/1 | 1/1 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Plitidepsin 2.5 mg (N=2) | Group 1: Control (N=1) | Group 2: Plitidepsin 2.5 mg (N=11) | Group 2: Control (N=4) | Group 3: Plitidepsin 2.5 mg (N=1) | Group 3: Control (N=1) | Group 4: Plitidepsin 2.5 mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Candida pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Plitidepsin 2.5 mg (N=2) | Group 1: Control (N=1) | Group 2: Plitidepsin 2.5 mg (N=11) | Group 2: Control (N=4) | Group 3: Plitidepsin 2.5 mg (N=1) | Group 3: Control (N=1) | Group 4: Plitidepsin 2.5 mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 5 (7) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Slow speech (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (7) | 1 (2) | 0 (0) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vein disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT05705167/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT05705167/SAP_001.pdf